CLINICAL TRIAL: NCT00749242
Title: Prospective Randomized Study Comparing Balloon Kyphoplasty and Conservative Treatment in Acute Traumatic Vertebral Fractures, Types A1, A2, AND A3.1 According to the Magerl Classification (STIC 3)
Brief Title: Comparative Study of Balloon Kyphoplasty and Conservative Treatment
Acronym: TRAUMAA1-2-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060110
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2012-11

CONDITIONS: SPINAL Fracture
Keywords: Traumatic vertebral fracture; Vertebroplasty; Balloon kyphoplasty; Bohler bracing
MeSH Terms: conditions — Spinal Fractures | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): conventional orthopedic brace with antalgic treatment
  Interventions: Other: orthopedic brace
- 2 (Other): balloon kyphoplasty introduction of balloon into the vertebral body, inflation of the balloon which creates a cavity, then balloon is deflated and removed , then introduction of the cement into the cavity.
  Interventions: Device: balloon kyphoplasty

INTERVENTIONS:
Other: orthopedic brace — antalgic drugs and orthopedic brace
  Other Names: böhler brace
  Arms: 1
Device: balloon kyphoplasty — introduction of balloon into the vertebral body, inflation of the balloon which creates a cavity, then balloon is deflated and removed , then introduction of the cement into the cavity.
  Arms: 2

SUMMARY:
This study will compare two treatments in acute stable traumatic vertebral fractures (types A1, A2 and A3.1 in MAGERL Classification). The two treatments are the followings:

1. Conservative Orthopedic Management consisting of brace and pain medication.
2. Percutaneous Balloon Kyphoplasty, a variant of Vertebroplasty, in which a balloon is first placed into the fractured vertebra and inflated with fluid in order to create a cavity. This may restore part of the vertebral height loss due to the fracture and facilitate the injection of the cement with low pressure.

The primary outcome will be the variation in the angle of Regional Vertebral Kyphosis (or, in the case of asymmetrical fractures, the angle of lateral vertebral inclination) between inclusion and one year follow-up. It will indicate if Balloon Kyphoplasty is able to restore vertebral height of the fractured vertebra better than Conservative Orthopedic Management.

DETAILED DESCRIPTION:
There is no reported frequency of stable thoracic or lumbar fractures traumatic fractures. However, the number of cases has been evaluated to be 61,425 yearly in Europe. Types A1 and A3.1 represent 61% of this number i.e. 37,468 per year in Europe and 4,600 in France.Conventional Conservative treatment of these fractures consists of brace and pain medication. However, a growing number of surgical teams use vertebroplasty or Balloon Kyphoplasty to avoid secondary fracture displacement after brace removal which results in increased kyphosis. However no study has compared the benefit of these new techniques to conservative managementThe goal of this study is to indicate if balloon kyphoplasty is able to restore vertebral height of the fractured vertebra better than Conservative Treatment.

1. The conventional orthopedic treatment is based on The Böhler Brace which extends from the manubrium to the pubic symphysis allowing spinal immobilisation in position of lumbar lordosis. Patients wear it for 3 to 6 months. It is a non-invasive treatment. However, kyphotic spine angle may increase over time despite the brace due to spine loading .

2 . Balloon Kyphoplasty is a variant of vertebroplasty which is performed under general anaesthesia using the KyphX® System (Medtronic., Sunnyvale, California). Balloon kyphoplasty aims at restore vertebral height of the fractured vertebra using an inflatable balloon prior to inject surgical cement (PMMA) into the vertebral body to fix the fracture. It is an expensive technique costing around 4,000 euros for up to 2 vertebrae in the same patient. The surgical technique for the procedure has been described by Lieberman and al: A bilateral approach is chosen to insert working cannulas into the posterior part of the vertebral body through a posterior transpedicular approach. Fluoroscopy is used to insert the tools and control the procedure. With reaming tools, two working channels are created and the balloons are inserted. The balloons are available in lengths of 10, 15 and 20 mm.The two balloons(one on each side) should ideally be centered at middle height between the superior and inferior endplates and in the anterior two-thirds of the vertebral body. Balloon placement into the vertebral body is checked using radiopaque markers at the two extremities of the balloon. Once inserted, the balloons are inflated using visual, volume and pressure control to create a cavity. Inflation is stopped when one of the following inflation endpoints is reached: pressure raised over 400 psi, balloon contacts one of the cortical bone of the vertebra or reaching maximal balloon inflation volume. The balloons are then deflated and removed. The mean balloon inflation volume is 2 to 3ml. The Bone Filler Device, filled before with 1.5 ml of polymethylmethacrylate (PMMA), is then advanced through the working cannula towards the anterior part of the cavity and cement is slowly extruded by a stainless steel stylet, acting as a plunger. When the amount of cement from the first Bone Filler Device is delivered in the cavity, it is removed and another Bone Filler Device is advanced through the working cannula. This step is repeated till a complete fill of the cavity is obtained. The same procedure is repeated through the other working cannula at the contra-lateral pedicle. Filling of the cavity with highly viscous PMMA is performed under continuous fluoroscopic control.

ELIGIBILITY:
Inclusion Criteria:

* Preliminary clinical exam (the anesthetist must have provided his approval for the surgical procedure)
* Patient must have signed the consent form (ZELEN Randomization protocol)
* Male or Female, 18 years or older;
* One to three traumatic fractures, non pathological, painful, less than 10 days of age, between T11 and L5 MAGERL A1 or A2 or A3.1. all the fractures should meet the inclusion criteria(deformity, aetiology, technical possibility of doing procedure). All fractures should received the same treatment
* Thoracic vertebral Kyphosis >15° or Lumbar vertebral Kyphosis > 10°, or Lateral angulation > 10°.
* Pain with VAS ≥ 5.
* The benign nature of the vertebral fracture has to be confirmed by the results of the biopsy performed during balloon kyphoplasty, or by one year follow-up in the Böhler Brace Group.
* Technical feasibility of a balloon kyphoplasty and Bohler bracing within 7 days after patient randomization.

Exclusion Criteria:

* Vertebral fracture of more than 10 day duration
* Vertebral fracture not located between T11 and L5
* Vertebral fracture type different from types A1, A2 and A3.1 according to MAGERL classification.
* Thoracic vertebral Kyphosis ≤ 15° or Lumbar vertebral Kyphosis ≤ 10°, or Lateral angulation ≤ 10°.
* Osteoporotic vertebral fracture
* Association to other post traumatic fractures.
* Neurological signs or symptoms related to the vertebral fracture
* History of spine fracture, kyphoplasty, spine surgery at thoracic or lumbar levels with low back pain.

History of surgery is not per sue a contraindication if there is no residual low back pain. However, in case of spinal fusion history, the fracture to be treated should be at minimum of two disc space from the most proximal or distal end of the fusion.

* Current infection
* Impossibility to perform the percutaneous approach of the vertebra to treat.
* Known allergy to the contrast product used during the Kyphoplasty procedure or to any of the cement components
* Reduction by more than 50% of the anteroposterior width of the bony spinal canal due to the vertebral fracture to treat.
* Vertebral fracture with loss of 90% or more of the vertebral body height
* Malignant and traumatic vertebral fractures
* Contraindication to MRI :

Metallic implant : pacemaker, non-movable auditive implant, metallic vascular or cardiac device Metallic surgical clips Claustrophobia

* Evolutive cardiac disease nonreactive to medical treatment
* Patient presenting a non correctable spontaneous or therapeutic coagulation disorder.
* Non compliant patient: Impossibility to participate to the study and to be followed up for 1 year.
* Pregnant or breast feeding women
* Patient not affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the variation of the angle of Vertebral Kyphosis or, in the case of asymmetrical fractures, the angle of lateral vertebral inclination between inclusion and one year follow-up examination | 1 year

SECONDARY OUTCOMES:
Pain evaluation using a visual analogic scale | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
questionnaire for back pain evaluation : Eifel | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Quality of life evaluation (SF 12). | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Analgesics intake according to the WHO classification (Classes 1, 2 and 3). | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Regional spine Kyphosis angle and global thoracic and lumbar Kyphosis angle | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Changes in anterior, mid and posterior vertebral heights of the treated vertebral body | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Changes in height of the intervertebral disc spaces adjacent to the treated vertebra | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Number of new vertebral fractures occurring during the one year follow-up period. | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Cost evaluation in a sample of 10% of patients randomly selected including the following costs : o Intervention cost.o Medical treatment costs o Consultation costs. o Hospitalization cost o Complication costs | J-20 à J-7 / J6 / J45 /J90 /J180 / J360
Follow-up of anterior, median and posterior height of the treated vertebral body, obtained by making an average of all measurements, on 3 cuts tomodensitometry (TDM) on the sagittal level : lateral right, median and lateral left | preoperative, at J6 and at J360
Intensity of signal with T2 sequence | preoperative and at J360

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis LAREDO, MD, Pr, Principal Investigator — AP-HP Assistance Publique- Hôpitaux de Paris
Locations (1):
- Hopital LARIBOISIERE Service de Radiologie Ostéo-Articulaire, Paris, France